CLINICAL TRIAL: NCT07362511
Title: Imagery Rescripting Within Primary Care to Manage Depression: A Single-Case Experimental Design
Brief Title: Imagery Rescripting in Primary Care
Acronym: IMPACT MADE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Amsterdam (Other)
Collaborators: UvA Huisartsen (Unknown)
Responsible Party: Principal Investigator, Lotte Stemerding, Dr., University of Amsterdam
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMG-11030
Record Dates: First submitted 2025-12-16; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Major Depressive Diorder; Low Self-Esteem; Mood Disorders
Keywords: Imagery Rescripting; Depression; Primary care
MeSH Terms: conditions — Mood Disorders; Depression

STUDY DESIGN:
Intervention Model Description: A multiple-baseline case series design will be used. All participants will first complete a baseline phase without intervention, and then undergo 10 weeks of Imagery Rescripting intervention (5 sessions). Participants are randomized to different waitlist (baseline) durations (2, 3 or 4 weeks), and intervention effectiveness is evaluated by comparing the change over time of bi-weekly self-reported depressive symptoms, self-esteem, and core beliefs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Imagery Rescripting (Experimental): The ImRs will follow the protocol as developed by Arntz and Weertman (1999), that was tailored for the primary care setting. The total of sessions will be set at 6. In session 1, the patient and therapist will create a list of core beliefs and memories to be rescripted. Session 1 will take place before the baseline phase, allowing us to assess core beliefs prior to the intervention. In session 2-6, one negative emotional memory is selected and rescripted (45 minutes per session). If necessary, a memory can be rescripted twice. In session 2-3 the therapist enters the image and rescripts the memory, whereas in session 4-6 the patient adult-self enters the image and rescripts the memory. If patients are uncomfortable doing so, session 4 can still be guided by the therapist.
  Interventions: Behavioral: Imagery Rescripting

INTERVENTIONS:
Behavioral: Imagery Rescripting — During ImRs, the patient brings a negative memory to mind and changes, together with the therapist, the outcome of the memory into a more positive
  Other Names: ImRs

SUMMARY:
In the current study we aim to investigate the feasibility, acceptability, and effectiveness of ImRs offered by mental health assistants within primary care to reduce depressive symptoms. In a single-case experimental design (SCED) study, the following hypotheses will be tested:

1. ImRs results in a reduction of depressive symptoms compared to baseline, and this reduction lasts up to six months.
2. Patients with complaints of depressive symptoms find ImRs an acceptable form of intervention when offered by mental health assistants within a general practice setting.

Participants will wait for 2-4 weeks and then receive 5 sessions of ImRs over a period of 10 weeks. During these sessions, negative memories related to their depressed feelings are rescripted.

DETAILED DESCRIPTION:
The study consists of a multiple-baseline case series in which the effectiveness and feasibility of Imagery Rescripting as a therapeutic technique will be investigated within primary care, with the aim of reducing depressive symptoms. The intervention will be provided by the mental health assistants (POH-GGZ) at the GP practice that is linked to the University of Amsterdam (Huisartsenpraktijk UvA). These mental health assistant have been trained in Imagery Rescripting. In the study, participants are randomly assigned to a baseline condition of 2-4 weeks, and a subsequent intervention condition of 10 weeks. During the intervention, all patients receive five sessions of Imagery Rescripting (45 minutes per session). Throughout these 12-14 weeks, and for 4 weeks after, participants complete bi-weekly (i.e., twice per week) measurements. The total number of bi-weekly measurements is thus 32-36, depending on the baseline condition that participants are randomized to. In addition, there will be 5 longer questionnaires, including a 3 and 6-month follow-up. Participants that are invited to the study but that do not want to participate will receive care as usual by the mental health assistant.

ELIGIBILITY:
Inclusion Criteria:

* Main complaint of depressive feelings, as indicated by both the mental health assistant and the patient.
* HADS score for the depression subscale ≥ 11.
* Ability to understand, read, write and speak Dutch or English.
* Age between 18 and 70.
* Willingness to participate in the study and treatment.

Exclusion Criteria:

* Acute suicide risk (BDI-II-item9 score of 3).
* If the mental health assistant suspects that the patient may have a primary diagnosis of bipolar disorder, psychosis, substance use disorder, low IQ, or if the patient suffers from serious neurological problems such as dementia, then the patient is not included. There will not be a formal assessment of a primary diagnosis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Depressive symptom severity | 16-18 weeks, twice a week
  Depressive symptom severity is assessed with the PHQ-2 (Kroenke et al., 2003). The PHQ-2 consists of the first two items of the PHQ-9 and measures the frequency of depressed mood and anhedonia in the past week. Scores range from 0-6 and higher scores mean more depressive symptoms.
Self-esteem | 16-18 weeks, twice a week
  Self-esteem will be measured with a single question "How have you felt about yourself in the past week?" Participants rate this question on a scale from -100 (very negative) to +100 (very positive).
Dysfunctional core beliefs | 16-18 weeks, twice a week + 3 month and 6 month follow-up
  Participants will formulate these negative beliefs about themselves or the world/other people together with the mental health assistant during the first session and then rate how convincing these beliefs are on a scale from 0 (not at all convincing) -100 (very convincing).

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale | Baseline, pre-treatment, 4-weeks post-treatment, 3 month follow-up, 6 month follow-up
  Measures depressive and anxious symptoms on a 14 item scale (Zigmond & Snaith, 1983). Scores range from 0-21 per scale (Anxiety and Depression) and higher scores reflect higher symptom severity.
Rosenberg Self-Esteem Scale | Baseline, pre-treatment, 4-weeks post-treatment, 3 month follow-up, 6 month follow-up
  Measures self-esteem with 10 items scored on a 4-point scale, scores range from 0 to 30, and higher scores reflect higher self-esteem (Rosenberg, 1965).
Suicidal thoughts | Baseline, pre-treatment, 4-weeks post-treatment, 3 month follow-up, 6 month follow-up
  Suicidal thoughts are measured using item 9 of Beck's depression inventory (BDI-II)
Emotional memory | Pre-treatment, 4-weeks post-treatment, 3 month follow-up, 6 month follow-up
  We will measure the following characteristics of the reported memories that will be rescripted: Vividness, Emotional Intensity, Emotional Impact, Intrusivity.
  These characteristics will be assessed with subscales of the Memory Experiences Questionnaire (MEQ; Vividness and Emotional Intensity) and two added subscales (Emotional Impact, Intrusivity). These measures are based on a previous study that these indices of a negative emotional memory related to depression scores (Stemerding et al., 2025). Each aspects is scored from 1-5 and higher scores mean stronger vividness, emotional intensity, emotional impact and intrusiveness.

OTHER OUTCOMES:
Acceptability | 4- weeks post-treatment
  We assess the acceptibility of the intervention using six questions that are formulated to measure how the participants feel about the intervention. An example is "To what extent would you recommend this intervention to a friend or family member that experiences symptoms similar to yours?". These items are assessed on a 9 point likert scale ranging from "not at all" to "very much".

CONTACTS AND LOCATIONS:
Locations (1):
- UvA Huisartsen, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
Due to privacy regulations we are not allowed to share individual patient data.